CLINICAL TRIAL: NCT06664918
Title: Effectiveness and Safety of the 4-Step Versus 6-Step Milk Ladder in Children with IgE-Mediated Cow's Milk Protein Allergy: Protocol for an Open-Label Randomised Controlled Trial
Brief Title: Effectiveness and Safety of Milk Ladders in Children with IgE-Mediated Cow's Milk Protein Allergy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrea Horvath-Stolarczyk, Associate Professor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML2024
Record Dates: First submitted 2024-10-16; First posted 2024-10-30 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cow Milk Allergy; Food Allergy
Keywords: IgE-mediated cow's milk allergy; children; milk ladder
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-step milk ladder (Experimental)
  Interventions: Other: oral food challenge (OFC)
- 6-step milk ladder (Active Comparator)
  Interventions: Other: oral food challenge (OFC)

INTERVENTIONS:
Other: oral food challenge (OFC) — oral food challenges with subsequent steps of 4-step milk ladder (muffin, pancake,baked hard cheese, yoghurt/pasteurised cow milk or modified cow milk)
  Arms: 4-step milk ladder
Other: oral food challenge (OFC) — oral food challenges with subsequent steps of 6-step milk ladder (cookie, muffin, pancake,baked hard cheese, yoghurt, pasteurised cow milk or modified cow milk)
  Arms: 6-step milk ladder

SUMMARY:
Cow's milk protein allergy (CMPA) is one of the most common food allergies in early childhood. The first-line treatment of CMPA is the elimination of cow's milk proteins (CMPs) from the child's or maternal diet.

Available data from the literature indicate that most children with CMPA acquire tolerance to CMPs with age. An assessment of tolerance acquisition to CMPs is commonly performed using milk ladder. However, scientific evidence regarding the effectiveness and safety of the milk ladder in children with CMPA is limited. Currently, there is no standardised milk ladder protocol, and different versions of the ladder and recommend by scientific societies in various countries.

This study aims to assess the effectiveness and safety of the 4-step milk ladder (4-ML) compared to the 6-step milk ladder (6-ML) in children with IgE-mediated CMPA. This is an open-label, randomised superiority trial with two parallel arms and a 1:1 allocation ratio.

DETAILED DESCRIPTION:
Introducing baked milk into the diet of children with cow's milk protein allergy (CMPA) has been shown to potentially accelerate the development of tolerance to raw milk. However, there is no standardised milk ladder protocol, and different scientific societies across countries recommend varying versions.

This study aims to assess the effectiveness and safety of the 4-step milk ladder (4-ML) compared to the 6-step milk ladder (6-ML) in children with IgE-mediated CMPA.

We will perform an open-label randomised trial with two parallel arms in two departments of the same academic hospital. A total of 92 children with IgE-mediated CMPA will be allocated to introduce cow's milk into their diet according to either 4-ML or 6-ML with a 4-week break period between subsequent steps. Oral food challenge (OFCs) with tested products at each subsequent step of the milk ladder will be conducted in hospital settings. The primary outcome will be the percentage of children with tolerance to non-heated cow's milk proteins defined as no allergic reaction to non-heated cow's milk (120-240 ml depending on the age of the patient) during the last OFC; measured at the end of the 12-week observation period for the 4-ML and 20-week observation period for the 6-ML. Secondary outcomes will include the percentage of children with a negative OFC to each milk ladder step; the percentage of children with anaphylaxis (both those who were treated and who were not treated with adrenaline); the percentage of children with exacerbation of atopic dermatitis; growth; compliance; and quality of life of the caregivers and parents' anxiety about adverse events during their child's OFC.

The statistical analyses will be conducted with StatsDirect. The Mann-Whitney U test will be used to compare the means of continuous variables if non-normal distribution will be assessed. Proportions will be compared with the Fisher exact test. The difference in study groups was considered significant when the P value will be <05. The results of this study will be analyzed on the basis of intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 5 years.
* Diagnosis of IgE-mediated CMPA confirmed according to ESPGHAN guidelines, by a positive OFC with CMPs. In high-risk children (i.e., with a history of anaphylaxis), diagnosis based on positive skin prick testing and/or elevated specific IgE to CMPs is sufficient.
* On a therapeutic elimination diet for at least 6 months or up to 12 months of age.12
* Eligible regardless of the risk of systemic reaction (anaphylaxis) and asthma.
* Good overall health status.
* Parents without language barriers.
* Written informed consent signed by parents.
* Good cooperation with the child's guardians.

Exclusion Criteria:

* Uncontrolled asthma, defined as the presence of shortness of breath, chest tightness, cough, and/or auscultatory changes despite treatment.
* Signs of exacerbation of a chronic disease.
* Signs of acute infectious disease (i.e., acute runny nose, cough, subfebrile fever, or fever).
* Signs of exacerbation of another allergic disease (i.e., conjunctivitis, allergic rhinitis, atopic dermatitis).
* Anaphylaxis due to CMPs in the last 6 months.
* Used antihistamines within 3-10 days before the challenge (depending on the characteristics of the drug and the reason for use).
* Acquired tolerance to baked CMPs or higher steps of the milk ladder.
* Use of immunosuppressive drugs or immunotherapy

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
The percentage of children who acquired tolerance to non-heated cow's milk proteins | at the end of the observation period (12 or 20 weeks, depending on the study arm)
  The percentage of children who acquired tolerance to non-heated cow's milk proteins defined as unreactive patients during OFC with non-heated cow's milk (the last step of milk ladder; a pasteurised cow milk or modified cow milk, the amount of 120-240 ml depending on the age of the patient, max. 7.95 g of CMPs)

SECONDARY OUTCOMES:
Percentage of children who experienced anaphylaxis | during the observation period (12 or 20 weeks, depending on the study arm)
  Anaphylaxis defined by the clinical criteria of anaphylaxis according to WAO 2020.
Percentage of children who required adrenaline administration | during the observation period (12 or 20 weeks, depending on the study arm)
Change in BMI-for-age z-score | at the end of the observation period (12 or 20 weeks, depending on the study arm) compared to baseline (before the first OFC)
Assessment of parents' anxiety about adverse events during their child's OFC | before each OFC, which means before the first OFC and depending on the study arm: after 4,8,12 weeks or after 4,8,12,16,20 weeks
  using the Subjective Units of Distress Scale (SUDS); parents will rate their level of anxiety on a scale from 1 to 100, where 0 represents no anxiety or complete relaxation, and 100 represents extreme anxiety, the worst ever experienced.
In a subgroup of children with atopic dermatitis, the percentage of children with mild, moderate, and severe atopic dermatitis | before and after each OFC (during the examination following each observation period) which means before and after the first OFC and and before and after subsequent OFCs depending on the study arm: after 4,8,12 weeks or after 4,8,12,16,20 weeks
  assessed using the oSCORAD23 scale; the maximum score on this scale is 83 points (in the most severe cases, an additional 10 points can be added for changes that disfigure or limit the patient's functioning), the minimum score is 0 points; the more points, the greater intensity of changes
Percentage of children with full compliance to the intervention protocol | at the end of the observation period (12 or 20 weeks, depending on the study arm)
  defined as performing all OFCs in the hospital setting and then regular introduction of the milk-containing products according to the individual tolerance following the Study Protocol
Percentage of children with negative OFCs to each cow's milk form after receiving the full planned amount for each OFC | at the end of the observation period (12 or 20 weeks, depending on the study arm)
  This will be reported as a percentage of children with negative OFCs to each cow's milk form (cookie, muffin, pancake, cheese, yoghurt, milk, if applicable) according to the milk ladder protocol, after receiving the full planned amount for each OFC.
Percentage of children with negative OFCs to each cow's milk form after receiving any tolerated dose | after the end of the observation period (12 or 20 weeks, depending on the study arm)
  This will be reported as a percentage of children with negative OFCs to each cow's milk form (cookie, muffin, pancake, cheese, yoghurt, milk, if applicable) according to the milk ladder protocol, after receiving any tolerated dose during the trial.
Change in total score of The Food Allergy Questionnaire of Life - Parent Form (FAQLQ-PF) | at the end of the observation period (12 or 20 weeks, depending on the study arm) compared to baseline (before the first OFC)
  The questionnaire is divided into three domains: emotional impact, food anxiety, and social and dietary limitations. The total score is calculated as the mean of three subscales. The minimum score is 0, the maximum score is 6. The lower the score, the more life affecting the allergy is.
Change in length/height-for-age z-score | at the end of the observation period (12 or 20 weeks, depending on the study arm) compared to baseline (before the first OFC)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Horvath, Principal Investigator — Medical University od Warsaw; Hanna Szajewska, Principal Investigator — Medical University of Warsaw; Anna Nowak-Węgrzyn, Principal Investigator — Collegium Medicum, University of Warmia and Mazury, Olsztyn, Poland; New York Univeristy, Grossmann School of Medicine
Locations (2):
- Poland (2):
  - Medical University od Warsaw, Department od Pediatrics, Warsaw
  - Medical University od Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
The results of this RCT, whether positive or negative, will be published in a peer-reviewed journal (data will be submitted to the first journal after 3-6 months from study completion). Abstracts will also be submitted to relevant national and international conferences.
  The datasets used and/or generated during this study will be made available from a given author upon reasonable request, after the publication of results, no later than 3 years from the completion of data analysis.
Supporting Information: Study Protocol
Time Frame: After the publication of results, no later than 3 years from the completion of data analysis with no end date.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Derived] Wiszniewska D, Horvath A, Strozyk A, Nowak-Wegrzyn A, Grzela K, Szajewska H. Effectiveness and safety of the four-step versus six-step milk ladder in children with IgE-mediated cow's milk protein allergy: protocol for an open-label randomised controlled trial. BMJ Open. 2025 Apr 14;15(4):e098314. doi: 10.1136/bmjopen-2024-098314. PMID 40228856